CLINICAL TRIAL: NCT01210885
Title: Phase 2, Observer Blinded, Controlled, Randomized Multi-Center Study in Adolescents, to Evaluate Safety, Tolerability and Immunogenicity of Four Different rMenB Plus MenACWY Formulations
Brief Title: Immunogenicity and Safety of Different rMenB Plus MenACWY Formulations in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V102_02
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal Disease; Vaccines; Adolescents
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (6):
- Group I: Investigational MenABCWY Formulation 1 (Experimental)
  Interventions: Biological: Meningococcal Vaccine
- Group II: Investigational MenABCWY Formulation 2 (Experimental)
  Interventions: Biological: Meningococcal Vaccine
- Group III: Investigational MenABCWY Formulation 3 (Experimental)
  Interventions: Biological: Meningococcal Vaccine
- Group IV: Investigational MenABCWY Formulation 4 (Experimental)
  Interventions: Biological: Meningococcal Vaccine
- Group V: Active comparator investigational MenB (Active Comparator)
  Interventions: Biological: Meningococcal Vaccine
- Group VI: Active comparator MenACWY (Active Comparator)
  Interventions: Biological: Meningococcal Vaccine

INTERVENTIONS:
Biological: Meningococcal Vaccine — MenABCWY combination vaccine containing four different rMenB formulations with MenACWY, intramuscular (IM) administration, vaccination at 0 and 2 months.

SUMMARY:
The purpose of this phase 2 study is to evaluate the safety, tolerability and immunogenicity of two doses of 4 different investigational MenABCWY combination vaccine when administered to healthy adolescents aged 11-18 years.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to be enrolled into this study are male and female subjects:

1. 11-18 years at the time of enrollment;
2. who have given their written consent/assent and whose parents or legal guardians have given written informed consent at the time of enrollment;
3. who are available for all the visits scheduled in the study (i.e., not planning to leave the area before the end of the study period);
4. in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. History of any meningococcal vaccine administration;
2. Current or previous, confirmed or suspected disease caused by N. meningitidis;
3. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment;
4. Significant acute or chronic infection within the previous 7 days or fever (defined as temperature 38C) within the previous 3 days;
5. Antibiotics within 7 days prior to enrollment;
6. Pregnancy or nursing (breastfeeding) mothers;
7. Females of childbearing age who have not used or do not plan to use acceptable birth control measures, for the duration of the study. Oral, injected or implanted hormonal contraceptive, barrier methods (condom or diaphragm with spermicide), intrauterine device or sexual abstinence are considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods at least two months prior to study entry;
8. Any serious chronic or progressive disease (e.g., neoplasm, diabetes, cardiac disease, hepatic disease, progressive neurological disease or seizure disorder; autoimmune disease, human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition);
9. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, including use of corticosteroids in immunosuppressive doses or chronic use of inhaled high-potency corticosteroids within the previous 60 days. [Use of topical corticosteroids administered during the study in limited areas (i.e., eczema on knees or face or elbows) of the body is allowed]; immunostimulants;
10. Receipt of blood, blood products and/or plasma derivatives, or a parenteral immunoglobulin preparation within the previous 90 days;
11. History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component;
12. Individuals who received any other vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccines;
13. Individuals participating in any clinical trial with another investigational product 30 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study;
14. Individuals who are part of study personnel or close family members conducting this study;
15. Individuals with medical history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study;
16. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 495 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Serum Bactericidal Assay (SBA) Geometric Mean Titers (GMTs) | 3 months
Percentage of subjects with seroresponse, and human Serum Bactericidal Activity (hSBA) titer ≥ 1:8 and hSBA titer ≥ 1:4 to Neisseria meningitidis serogroups A, C, W-135 and Y | 3 months
Percentage of subjects with hSBA titer ≥ 1:5 to N. meningitidis serogroup B strains | 3 months
Number of participants with solicited local and systemic reactions | within 7 days after each vaccination
Number of participants with any adverse events (AEs) | 6 months
Number of participants with Serious Adverse Events (SAEs) | 3 months

CONTACTS AND LOCATIONS:
Locations (8):
- Chile (3):
  - CESFAM Gabriela Mistral, Santiago
  - Liceo Carmela Carvajal de Prat, Santiago
  - Pontificia Universidad Católica de Chile, Santiago
- Colombia (3):
  - CafeSalud M P (Dir. de Investigación y Proyectos Especiales), Bogotá
  - Centro de Atencion e Investigacion Medica - CAIMED, Bogotá
  - Centro de Investigaciones CAFAM, Bogotá
- Panama (2):
  - Health Research International, Panama City
  - Indicasat, Panama City

REFERENCES:
- [Derived] Saez-Llorens X, Aguilera Vaca DC, Abarca K, Maho E, Grana MG, Heijnen E, Smolenov I, Dull PM. Immunogenicity and safety of investigational vaccine formulations against meningococcal serogroups A, B, C, W, and Y in healthy adolescents. Hum Vaccin Immunother. 2015;11(6):1507-17. doi: 10.1080/21645515.2015.1029686. PMID 25969894